CLINICAL TRIAL: NCT03689322
Title: Effects of Whole Body Vibration Associated With the Inspiratory Muscle Training Program on Inflammatory Markers, Body Composition, Muscle Strength and Thickness
Brief Title: Effects of WBV Associated With IMT on Inflammatory Markers, Body Composition, Muscle Strength and Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helga Cecília Muniz de Souza, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WBV on inflammatory biomarkers
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Frail Elderly Syndrome
Keywords: aging; whole body vibration; respiratory muscle training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WBV + IMT (Experimental): Whole body vibration training associated with respiratory muscle training (WBV + IMT)
  Interventions: Other: WBV + IMT
- WBV + IMTsham (Active Comparator): Whole body vibration training associated with respiratory muscle training sham (WBV + IMTsham)
  Interventions: Other: WBV + IMTsham
- WBVsham + IMTsham (Sham Comparator): Whole body vibration training sham associated with respiratory muscle training sham (WBVsham + IMTsham)
  Interventions: Other: WBVsham + IMTsham

INTERVENTIONS:
Other: WBV + IMT — The whole body vibration training will be performed through a vibrating platform with three axes and vibration frequency set at 35 Hz. The amplitude used will be 02 to 04 mm.The inspiratory muscle training will be performed through a device that provides inspiratory resistance.
  Arms: WBV + IMT
Other: WBV + IMTsham — The whole body vibration training will be performed through a vibrating platform with three axes and vibration frequency set at 35 Hz. The amplitude used will be 02 to 04 mm.The inspiratory muscle training sham will be performed through a device without inspiratory resistance.
  Arms: WBV + IMTsham
Other: WBVsham + IMTsham — Whole body vibration training will be performed through a vibrating platform coupled to a device that generates non-therapeutic low frequency vibration. The simulation of inspiratory muscle training will be performed through a device with no inspiratory resistance.
  Arms: WBVsham + IMTsham

SUMMARY:
Aging generates immune, muscular and functional changes. In the pre-frail elderly these changes may be increased and, therefore, preventive interventions are indicated to minimize the consequences of sarcopenia in this population. This study aims to evaluate the effects of a whole body vibration training associated with the training of inspiratory muscles on the inflammatory, muscular and body composition outcomes in pre-frail elderly women.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals able to walk without assistance
* Good understanding to carry out the proposed tests, evaluated through the Mini Mental State Examination (MMSE).

Exclusion Criteria:

* Contraindication or difficulty to perform evaluation procedures
* Users of medications that interfere with the cardiovascular and / or muscular system
* Smokers
* Neuromuscular or degenerative diseases
* Pulmonary comorbidities
* Heart diseases
* Labyrinthitis.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength and Resistance | Change from Baseline respiratory muscle strength and resistance at 3 months
  Maximum Inspiratory and Expiratory Pressure will be evaluated through manovacuometer

SECONDARY OUTCOMES:
Thickness of the quadriceps muscle | Change from Baseline thickness of the quadriceps muscle at 3 months
  Ultrasound will be used to assess the thickness of the quadriceps muscle according to the pre-established protocol.
Diaphragmatic thickness | Change from Baseline diaphragmatic thickness at 3 months
  Ultrasound will to use to evaluate diaphragm thickness non-invasively in the zone of apposition during tidal breathing and with changes in lung volume.
Diaphragmatic mobility | Change from Baseline diaphragmatic mobility at 3 months
  During respiration to total lung capacity, measurement of the diaphragmatic excursion will be assessed by ultrasonography.
Body Composition | Change from Baseline body composition at 3 months
  Body composition will be evaluated through bioimpedance balance
Inflammatory markers | Change from Baseline inflammatory markers at 3 months
  Blood concentration of Interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha) and brain-derived neurotrophic factor (BDNF) will be assessed through blood plasma sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil